CLINICAL TRIAL: NCT02138240
Title: Sugar Champ: Pilot Social Network Intervention to Reduce Intake of Sugary Drinks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00107116; K23HL116601 (NIH)
Record Dates: First submitted 2014-05-09; First posted 2014-05-14 (Estimated); Results first posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-06

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Social network intervention (Experimental): Individuals will be recruited and trained to be "Peer Educators" who will participate in group sessions and then communicate this information with members of participant's social network ("Sidekick") and work to make changes to reduce intake of sugar-sweetened beverages. Peer Educators will participate in 6 core group sessions over a 6-week period as well as 3 additional booster sessions over the subsequent 3 months after completing the core curriculum. All sessions will be delivered by a facilitator and assistant facilitator using a guide.
  Interventions: Behavioral: Social network intervention

INTERVENTIONS:
Behavioral: Social network intervention — The intervention combined a social network approach with strategies that address public housing residents' challenges related to the built environment to improve dietary habits. Given the frequent intake of sugar-sweetened beverages (SSB) in this population, the intervention focused on reducing added sugar intake through the reduced consumption of SSB.

SUMMARY:
The 1.2 million households living in public housing are disproportionately affected by obesity, where prevalence is estimated at 50%. An ecologic framework hypothesizes that this disparity is related, in part, to social and environmental factors within these neighborhoods that influence residents' lifestyles. Social networks and the built environment may work together to promote or inhibit lifestyle behaviors; however, combined social network-built environment interventions have not previously targeted changes in diet. Investigators hypothesize that an intervention that combines a social network approach with strategies that address public housing residents' challenges related to the built environment will improve dietary habits. The investigators' overall aim is to develop a combined social network-built environment intervention to reduce intake of beverages high in added sugars and to pilot test the intervention among residents of public housing developments in Baltimore, MD. The investigators' aim for this work is: 1) To develop a combined social network-built environment intervention to reduce intake of beverages high in added sugars and to pilot test the intervention among residents of public housing developments in Baltimore, MD. Investigators hypothesize that a social network intervention will be feasible and acceptable in promoting healthy lifestyle change, and that this intervention will alter lifestyle behaviors among public housing residents.

DETAILED DESCRIPTION:
Investigators will conduct a 6-month non-randomized trial of the social network intervention described below. This will be a single arm trial in which investigators compare the outcomes of interest pre- and post- intervention. Investigators will adapt an HIV risk reduction social network intervention to create a new social network intervention targeting reduction in intake of sugar-sweetened beverages (SSB). The investigators' primary outcomes will be to test the acceptability and feasibility of the intervention and its components as well as estimate the likely effect of the intervention.

In the intervention, individuals will be recruited and trained to be "Peer Educators" who will participate in group sessions and then communicate this information with members of participant's social network ("Sidekick") and work to make changes to reduce intake of added sugars together. Given the frequent intake of SSB in this population, the intervention will focus on reducing added sugar intake through the reduced consumption of SSB. Peer Educators will participate in 6 core group sessions over a 6-week period as well as 3 additional booster sessions after completing the core curriculum. All sessions will be delivered by a facilitator and assistant facilitator using a guide. All groups will be held in a room in each public housing development's administrative building.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* BMI≥25 kg/m2
* Must consume sugar-sweetened beverages at least twice daily
* "Peer Educators" must identify one high-risk alter in the social network to enroll as "Sidekick"
* Resides in select public housing developments in Baltimore, MD

Exclusion Criteria:

* Any underlying medical conditions that could seriously reduce life expectancy, ability to participate in the trial, or for which lifestyle change may be contraindicated and/or require medical supervision by a physician such as medication-dependent diabetes mellitus, cancer, lung disease requiring supplemental oxygen, dementia, angina, or diagnosis in the last 12 months of myocardial infarction, transient ischemic attack or stroke
* Women who are pregnant or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Gudzune, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Social Network Intervention: Individuals will be recruited and trained to be "Peer Educators" who will participate in group sessions and then communicate this information with members of their social network ("Sidekick") and work to make changes to reduce intake of sugar-sweetened beverages. Peer Educators will participate in 6 core group sessions over a 6-week period as well as 3 additional booster sessions over the subsequent 3 months after completing the core curriculum. All sessions will be delivered by a facilitator and assistant facilitator using a guide.
  Social network intervention: The intervention combined a social network approach with strategies that address public housing residents' challenges related to the built environment to improve dietary habits. Given the frequent intake of sugar-sweetened beverages (SSB) in this population, the intervention focused on reducing added sugar intake through the reduced consumption of SSB.
Period: Overall Study
Arm/Group | Social Network Intervention
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Social Network Intervention
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African-American | 33
  Other | 1
Added sugar intake total sample [Median (Inter-Quartile Range); unit: teaspoons/day] — Participants answered questions from the National Health Interview Survey (NHIS) 5-factor dietary screener. Relevant elements as recommended by NHIS were combined to estimate the daily added sugar intake (i.e.,soda, sugar-sweetened beverages, sweets and doughnuts). Prior assessments of African-Americans report that typical added sugar intake is 13.9 and 19.4 teaspoons/day among women and men, respectively. The American Heart Association recommends that all adults limit their added sugar intake to no more than 9 teaspoons per day. Baseline range (min-max) in this sample 14.1-78.9 teaspoons/day.
  teaspoons/day | 38.0 [28.3 to 47.5]
Added Sugar Intake among Sidekicks [Median (Inter-Quartile Range); unit: teaspoons/day] — Participants answered questions from the National Health Interview Survey (NHIS) 5-factor dietary screener, and relevant elements as recommended by NHIS were combined to estimate the daily added sugar intake (i.e.,soda, sugar-sweetened beverages, sweets and doughnuts). Population: Limited to only Sidekicks
  teaspoons/day
    number analyzed (Participants) | 17
    (all) | 37.0 [30.8 to 41.1]
Added Sugar Intake among Peer Educators [Median (Inter-Quartile Range); unit: teaspoons/day] — Participants answered questions from the National Health Interview Survey (NHIS) 5-factor dietary screener, and relevant elements as recommended by NHIS were combined to estimate the daily added sugar intake (i.e.,soda, sugar-sweetened beverages, sweets and doughnuts). Population: Limited to only Peer Educators
  teaspoons/day
    number analyzed (Participants) | 17
    (all) | 42.4 [18.4 to 57.6]
Weight, continuous [Median (Inter-Quartile Range); unit: kg] | 85.9 [73.5 to 96.9]
Body mass index, continuous [Mean (Standard Deviation); unit: kg/m^2] | 32.1 (6.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Sessions Attended
Description: Number of sessions attended calculated from attendance sign-in sheets. This is used for the assessment of program feasibility.
Time Frame: 3 months
Population: Limited to Peer Educators who had the opportunity to attend the sessions.
Measure: Median (Inter-Quartile Range); unit: Number of sessions
Arm/Group | Social Network Intervention
Number analyzed (Participants) | 17
Number of sessions | 9 [4 to 9]

2. Primary Outcome: Participant Satisfaction as Assessed by 4-point Likert Scale
Description: Survey question assesses participant satisfaction with the intervention using a 4-point Likert scale (1 = Very satisfied; 2= Somewhat satisfied; 3 = Somewhat dissatisfied; 4 = Very dissatisfied). This is used for the assessment of program acceptability.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Social Network Intervention
Number analyzed (Participants) | 34
Participants
  Very satisfied | 30
  Somewhat satisfied | 4
  Somewhat dissatisfied | 0
  Very dissatisfied | 0

3. Primary Outcome: Participant's Likelihood to Recommend Program Assessed by 4-point Likert Scale
Description: Survey question assesses willingness to recommend that a friend participate using a 4-point Likert scale (1 = Very likely; 2= Somewhat likely; 3 = Somewhat unlikely; 4 = Very unlikely). This is used to assess the program acceptability.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Social Network Intervention
Number analyzed (Participants) | 34
Participants
  Very likely | 31
  Somewhat likely | 3
  Somewhat unlikely | 0
  Very unlikely | 0

4. Primary Outcome: Added Sugar Intake (Teaspoons/Day) Among Total Sample at Follow up
Description: Participants answered questions from the National Health Interview Survey (NHIS) 5-factor dietary screener, and relevant elements as recommended by NHIS were combined to estimate the daily added sugar intake (i.e.,soda, sugar-sweetened beverages, sweets and doughnuts). At 6 months, this measure ranged (min-max) from 9.1 to 56.0 teaspoons/day in this sample. The American Heart Association recommends that all adults limit their added sugar intake to no more than 9 teaspoons per day.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: teaspoons/day
Arm/Group | Social Network Intervention
Number analyzed (Participants) | 34
teaspoons/day | 17.2 [11.2 to 27.8]
Statistical Analysis 1: Comparison: Social Network Intervention; Test type: Other — Pre-post comparison; p < 0.001, Wilcoxon signed rank sum

5. Secondary Outcome: Added Sugar Intake (Teaspoons/Day) Among Alters ("Sidekicks") at Follow up
Description: Participants answered questions from the National Health Interview Survey (NHIS) 5-factor dietary screener, and relevant elements as recommended by NHIS were combined to estimate the daily added sugar intake (i.e.,soda, sugar-sweetened beverages, sweets and doughnuts). The American Heart Association recommends that all adults limit their added sugar intake to no more than 9 teaspoons per day.
Time Frame: 6 months
Population: Limited to Sidekicks only
Measure: Median (Inter-Quartile Range); unit: teaspoons/day
Arm/Group | Social Network Intervention
Number analyzed (Participants) | 17
teaspoons/day | 16.9 [12.7 to 27.8]

6. Secondary Outcome: Added Sugar Intake (Teaspoons/Day) Among Egos ("Peer Educators") at Follow up
Description: as for outcome 5
Time Frame: 6 months
Population: Limited to Peer Educators
Measure: Median (Inter-Quartile Range); unit: teaspoons/day
Arm/Group | Social Network Intervention
Number analyzed (Participants) | 17
teaspoons/day | 17.4 [11.2 to 24.5]

7. Secondary Outcome: Median Weight at Follow up
Description: Weight (kg) measured using standard methods
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: kg
Arm/Group | Social Network Intervention
Number analyzed (Participants) | 34
kg | 84.3 [74.7 to 100.4]
Statistical Analysis 1: Comparison: Social Network Intervention; Test type: Other — Pre-post comparison of baseline median weight to median weight at 6-month follow up; p = 0.21, Wilcoxon signed rank sum

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Social Network Intervention
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-23): https://cdn.clinicaltrials.gov/large-docs/40/NCT02138240/Prot_SAP_000.pdf